CLINICAL TRIAL: NCT06990165
Title: Efficacy of Photobiomodulation in the Prevention and Severity of Radiodermatitis in People With Breast Cancer Undergoing Adjuvant Radiotherapy
Brief Title: Photobiomodulation in Radiodermatitis in People With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Anke Bergmann, Principal Investigator, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 83380324.4.0000.5274
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Radio Dermatitis
Keywords: Physical Therapy; Phototherapy; Low-Level Light Therapy; Radiodermatitis; Adverse effects; Radiotherapy Adjuvant; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomization will be by lot when the patient enters the study. Envelopes will be made available that will contain a code that determines the allocation of patients in the intervention group experimental or standard.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active photobiomodulation group (Group A) (Experimental): Will receive photobiomodulation using the Antares/IBRAMED® device with a cluster applicator, at two distinct wavelengths: infrared laser light (808 nm) and red light (630 nm).
  Interventions: Device: Photobiomodulation
- placebo photobiomodulation group (Group B) (Sham Comparator): Group B will undergo the same protocol as Group A, with the device making contact with the irradiated area, but the device will be turned off, therefore not emitting any therapeutic light.
  Interventions: Other: Sham Control

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation applications will be performed within 1 hour after the radiotherapy session, covering the entire irradiated area, three times per week, starting from the first day of radiotherapy. The procedure will be conducted using the Antares/IBRAMED® device, with a cluster applicator featuring a 20 cm² contact area and two distinct wavelengths: four infrared laser diodes (808 nm), each with a power of 180 mW, and three red light diodes (630 nm), each with a power of 150 mW. Each diode will deliver 3 J of energy, with the wavelengths applied separately and sequentially.
  Other Names: Low-Level Light Therapy; Photobiomodulation Therapy; Low-Level Laser Therapy; Low-Power Laser Irradiation; Laser Phototherapy
  Arms: active photobiomodulation group (Group A)
Other: Sham Control — Group B will have the device in contact with the irradiated area, following the same protocol as Group A, but with the device turned off, receiving no therapeutic light and, therefore, experiencing no biological effects from the light.
  Arms: placebo photobiomodulation group (Group B)

SUMMARY:
Most breast cancer patients undergoing radiotherapy develop radiodermatitis, making it one of the most prevalent adverse events during cancer treatment. The severity of radiodermatitis can pose a life-threatening risk to patients, lead to functional limitations, delay treatment (pauses for tissue recovery), reduce the radiation dose, and negatively impact health-related quality of life. There is no consensus on the ideal strategy for preventing radiodermatitis.

Photobiomodulation is a non-invasive strategythat may stimulate skin regeneration and minimize radiodermatitis without interfering with cancer treatment, with minimal risk (it may cause rare allergic-type complications or discomfort due to material contact) and low cost for both the patient and the healthcare system, making this approach highly relevant.

Reducing the use of pharmaceuticals, the duration of radiotherapy treatment, and the costs associated with managing radiodermatitis will have socioeconomic and environmental impacts, as this is a sustainable, safe, and cost-effective therapeutic approach with high applicability and clinical reproducibility.

Additionally, it can later be expanded to other types of cancer. This study hypothesizes that photobiomodulation can prevent and reduce complications associated with radiodermatitis in breast cancer patients undergoing adjuvant radiotherapy.

Therefore, the primary objective of this clinical trial is to assess the efficacy of photobiomodulation in preventing and reducing the severity of radiodermatitis in breast cancer patients receiving adjuvant radiotherapy at Hospital do Câncer III of the Brazilian National Cancer Institute.

The secondary objectives include evaluating the incidence and severity grades of radiodermatitis; comparing the influence of photobiomodulation, according to the intervention group, on the occurrence and severity of radiodermatitis, pain, edema/lymphedema, paresthesia, functionality, skin quality, health-related quality of life, and sleep quality after radiotherapy; comparing the recovery time of radiodermatitis between groups; and assessing satisfaction, safety, and tolerability of photobiomodulation use.

DETAILED DESCRIPTION:
This study is a Randomized Controlled Superiority Clinical Trial involving individuals diagnosed with breast cancer and indicated for adjuvant radiotherapy at Hospital do Câncer III of the National Cancer Institute (HCIII/INCA) in Rio de Janeiro. All individuals attending HCIII/INCA for their first consultation for adjuvant radiotherapy for breast cancer will be recruited to assess eligibility criteria for the study. Those deemed eligible will receive detailed explanations regarding the study objectives, treatment groups, adverse effects, and the voluntary nature of participation through the Informed Consent Form (ICF). Upon agreeing and signing the ICF, they will undergo an initial assessment and be randomized into one of the following groups: Active Photobiomodulation Group (intervention) or Placebo Photobiomodulation Group (control).

Randomization will follow a 1:1 allocation ratio between the two groups and will be conducted using sealed, opaque envelopes in blocks of ten patients, each containing an allocation code (five codes for Active Photobiomodulation Group and five codes for Placebo Photobiomodulation Group). This method was chosen to prevent biases related to therapist or participant preferences regarding the intervention. The participants will be informed about their assigned group and the follow-up procedures throughout radiotherapy and up to three months after treatment. All assessments, interventions, and data collection will be performed by trained and qualified professionals.

At the beginning of radiotherapy, all participants will receive guidance on skin care, specific home exercises for the upper limbs, and maintaining their usual physical activities, following the institutional standard of care.

Sociodemographic characteristics (age, race/skin color, education level, marital status, and per capita income) and clinical data (comorbidities, physical activity, tobacco and alcohol consumption, body mass index, physiotherapy follow-up, clinical staging, cancer treatment history, post-operative scar complications, and oncologic treatment-related complications) will be collected from physical and electronic medical records.

For data analysis, descriptive and comparative analyses will be performed between the intervention groups concerning selected variables and primary outcomes. Measures of central tendency and dispersion will be determined for continuous variables, and frequency distribution will be used for categorical variables. Outcome evaluations (primary and secondary) will follow an intention-to-treat analysis. The Kolmogorov-Smirnov test will be used to assess data normality. Chi-square tests will analyze categorical outcomes and will be presented in absolute and relative numbers. Student's t-tests will analyze parametric continuous outcomes and will be presented as mean and standard deviation, while the Mann-Whitney test will be used for non-parametric data, presented as median and minimum-maximum values. A significance level of p<0.05 and a 95% confidence interval will be considered for all analyses, which will be performed using SPSS (Statistical Package for the Social Sciences) version 24.

This research will not impose any financial burden on participants, as assessments will be conducted during routine consultations or treatment sessions, and additional data will be collected from electronic and/or physical medical records. The intervention materials (Antares photobiomodulation device by IBRAMED®, two protective glasses for the operator and patient, power cable, fuse, and operation manual) will be provided to the Clinical Epidemiology Applied to Oncology research group (on loan from IBRAMED® during the study period). Other office supply costs will be covered by the researchers responsible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older with an indication for adjuvant radiotherapy for breast cancer treatment at National Cancer Institute (INCA-BRAZIL).

Exclusion Criteria:

* Previous diagnosis of cancer or bilateral breast cancer.
* Oncological treatment outside the institution.
* Connective tissue disorders (such as scleroderma and lupus erythematosus).
* Previous radiotherapy to the breast or chest wall.
* Individuals unable to complete the questionnaires.
* Individuals unable to receive photobiomodulation due to acute infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of radiodermatitis as assessed by the Radiation Therapy Oncology Group / European Organisation for Research and Treatment of Cancer (RTOG/EORTC) Classification System over 5 months after the start of adjuvant radiotherapy. | Evaluations will be performed in baseline, once a week during treatment (which lasts an average of 5 weeks), as well as at 30 days and 3 months after the end of radiotherapy.
  The set of skin reactions caused by radiotherapy treatment is classified by the Radiation Therapy Oncology Group / European Organisation for Research and Treatment of Cancer (RTOG/EORTC) system as follows: Grade 0 - no reaction; Grade 1 - mild erythema, epilation, and dry desquamation; Grade 2 - painful erythema, moist desquamation, and moderate edema; Grade 3 - confluent moist desquamation and significant edema; Grade 4 - ulceration, hemorrhage, and necrosis.

SECONDARY OUTCOMES:
Incidence, intensity and modulation of pain assessed using the Visual Analog Scale (VAS) over 5 months after the start of adjuvant radiotherapy | Evaluations will be performed in baseline and each photobiomodulation intervention (which lasts an average of 5 weeks), as well as at 30 days and 3 months after the end of radiotherapy.
  Pain incidence, intensity and modulation will be assessed using the Visual Analog Scale (VAS) at each intervention. This is a Likert-type scale ranging from 0 (no pain) to 10 (unbearable pain).The VAS will be applied to each intervention, as well as at 30 days and 3 months after the end of radiotherapy.
Characteristics and intensity of pain assessed by the Pain DETECT questionnaire over 5 months after the start of adjuvant radiotherapy | Evaluations will be performed in baseline once a week during treatment (which lasts an average of 5 weeks), as well as at 30 days and 3 months after the end of radiotherapy.
  The Pain DETECT questionnaire is an instrument that characterizes the type of pain based on a score, which ranges from 1 to 38 points (≤ 12 points indicates an unlikely neuropathic component, with nociceptive pain; between 13 and 18 points, indicates mixed pain; and scores ≥ 19 points suggest a probable neuropathic component and neuropathic pain).
Pain components assessed by the McGILL questionnaire over 5 months after the start of adjuvant radiotherapy | Evaluations will be performed in baseline, once a week during treatment (which lasts an average of 5 weeks), as well as at 30 days and 3 months after the end of radiotherapy.
  The McGILL questionnaire is an instrument that characterizes the pain components as affective, sensory, and evaluativeproviding qualitative information through patient descriptions. The McGILL questionnair will be administered once per week during treatment, as well as at 30 days and 3 months after the end of radiotherapy.
Incidence and severity of edema/lymphedema over 5 months after the start of adjuvant radiotherapy. | Assessments will be conducted at the baseline and end of radiotherapy treatment, as well as at 30 days and 3 months after its completion.
  Assessments will be conducted at the beginning and end of radiotherapy, as well as at 30 days and 3 months after its completion, using upper limb perimetry. Measurement points will include: (1) elbow joint line (EJL); (2) 7 cm and 14 cm above the EJL; (3) 7 cm, 14 cm, and 21 cm below the EJL; and (4) the dorsum of the hand. The total limb volume will be calculated using the truncated cone formula based on circumference measurements:
  V = h * (C² + Cc + c²) / (π * 12), where 'V' represents the total segment volume of the limb, 'C' and 'c' are the circumferences at the measured points, and 'h' is the distance between the circumferences in each segment. Lymphedema will be defined as a total volume difference of ≥ 10% between the affected and contralateral limb after six months of surgical treatment. Edema will be defined as a total volume difference of ≥ 10% within the first six months after surgery.
Superficial sensitivity of the irradiated skin assessed by esthesiometry over 5 months after the start of adjuvant radiotherapy | Assessments will be conducted at the baseline and end of radiotherapy treatment, as well as at 30 days and 3 months after its completion.
  Assessments will be conducted at the beginning and end of radiotherapy, as well as at 30 days and 3 months after its completion, using an esthesiometer (monofilaments). The test will be demonstrated to the participant on an area of skin with normal sensitivity. The testing points will be predetermined, and the sequence of testing may be random. The test begins with the green filament (0.05g) at all points. If the participant does not feel the green filament at a given point, the blue filament is used, followed by the next in sequence if necessary. The participant will be asked to respond "yes" when they feel the touch. Each filament color, with its specific weight, represents a different sensitivity threshold, and the interpretation follows the manufacturer's manual recommendations.
Functionality of the upper limb on the irradiated side assessed by the Disability of Arm, Shoulder, and Hand (DASH) Questionnaire over 5 months after the start of adjuvant radiotherapy. | Evaluations will be performed in baseline , 30 days and 3 months after the end of radiotherapy.
  The Disability of Arm, Shoulder, and Hand (DASH) questionnaire is an instrument used to assess upper limb functionality. It consists of 30 questions and two optional modules. It uses a 5-point scale, with a total score ranging from 0 (no dysfunction) to 100 (severe dysfunction).
Skin quality over 5 months after the start of adjuvant radiotherapy, analyzed by thermography | The assessment will begin one week after the first radiotherapy session and will be repeated once a week during the treatment (which lasts on average 5 weeks), as well as 30 days and 3 months after the end of radiotherapy.
  Assessments will be conducted once per week during treatment, as well as at 30 days and 3 months after the end of radiotherapy, using a thermographic camera (which evaluates temperature and vascularization) and image analysis (pre- and post-intervention).
  The infrared thermographic camera will capture images, which will be processed using specialized software. Laboratory conditions will be controlled, maintaining an ambient temperature of 25.5±0.35°C and relative humidity of 50.5±2.16%. The camera will be positioned at an angle of approximately 90° to the surface and 1 meter from the participant to provide a complete view of the irradiated skin.
Health-Related Quality of Life assessed by the EORTC QLQ-C30 (3rd version) and EORTC QLQ-BR23 questionnaires over 5 months after the start of adjuvant radiotherapy. | Assessments will be conducted at the baseline and end of radiotherapy, as well as at 30 days and 3 months after its completion
  Assessments will be conducted at the beginning and end of radiotherapy, as well as at 30 days and 3 months after its completion, using two questionnaires developed by the European Organisation for Research and Treatment of Cancer (EORTC).
  The EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), 3rd version, is a multidimensional, self-administered questionnaire that includes 30 questions related to five functional scales, a global health status scale, and a symptom scale.
  The EORTC Quality of Life Questionnaire breast cancer module (EORTC QLQ-BR23) is a breast cancer-specific quality of life questionnaire containing 23 questions related to functional and symptom scales. These questionnaires have been translated and validated in Portuguese.
  Higher scores on functional scales indicate better quality of life, whereas higher scores on symptom scales represent poorer quality of life.
Sleep quality according to the Pittsburgh Sleep Quality Index (PSQI) over 5 months after the start of adjuvant radiotherapy | Assessments will be conducted at the baseline and end of radiotherapy, as well as at 30 days and 3 months after its completion
  The Pittsburgh Sleep Quality Index (PSQI) can be used for cancer patients and assesses sleep quality over a one-month period. It consists of seven components, each scored from 0 to 3, with a maximum total score of 21 points, where higher scores indicate poorer sleep quality.
  Scores above 5 points suggest poor sleep quality, distinguishing participants as "good sleepers" and "poor sleepers." The questionnaire will be administered at the beginning and end of radiotherapy, as well as at 30 days and 3 months after its completion.
Satisfaction and impact of photobiomodulation on participants' health condition at the end of radiotherapy | Approximately 5 weeks from the start of radiotherapy (21 days)
  The efficacy and overall satisfaction with the treatment of radiodermatitis, as well as the impact of the prevention and/or treatment of radiodermatitis with photobiomodulation on activities of daily living will be assessed at the end of radiotherapy through self-reporting of the incidence of adverse events emerging from treatment using a specific form.
Safety and tolerability to photobiomodulation | The assessment will begin one week after the first radiotherapy session and will be repeated once a week during the treatment (which lasts on average 5 weeks), as well as 30 days and 3 months after the end of radiotherapy.
  Assessment will be conducted once a week during treatment, as well as at 30 days and 3 months after the end of radiotherapy.
  The occurrence of adverse events related to photobiomodulation will be monitored to assess safety, and tolerability will be evaluated through participants' self-reports.
  Adverse events associated with the intervention will be assessed during follow-up evaluations using the Common Terminology Criteria for Adverse Events (CTCAE) and classified as Grade 1 (mild), Grade 2 (moderate), or Grade 3 (severe) including: Urticaria, pruritus, skin pain, eczema, dry skin and skin infection
Interruption of radiotherapy | Throughout radiotherapy
  It will be assessed by the responsible radiation oncologist. The date and reason for the interruption will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Bergmann, PhD, Principal Investigator — National Cancer Institute (INCA-BRAZIL)
Locations (2):
- Brazil (2):
  - National Cancer Institute (INCA-BRAZIL), Rio de Janeiro, Rio de Janeiro
  - National Cancer Institute / Cancer Hospital III - Brazil, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.